CLINICAL TRIAL: NCT00648648
Title: A Phase I Dose Escalation Study Evaluating MK-1775 in Both Monotherapy and in Combination With Either Gemcitabine, Cisplatin, or Carboplatin in Adult Subjects With Advanced Solid Tumors
Brief Title: A Dose Escalation Study of Adavosertib (MK-1775) in Combination With Either Gemcitabine, Cisplatin, or Carboplatin in Adults With Advanced Solid Tumors (MK-1775-001)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1775-001; 2007_611 (Other: Merck Registration Number); MK-1775-001 (Other: Merck Protocol Number); 2007-005304-40 (EudraCT Number)
Record Dates: First submitted 2008-03-26; First posted 2008-04-01 (Estimated); Results first posted 2019-04-05 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumors
MeSH Terms: interventions — adavosertib; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (28):
- adavosertib 325 mg Single Dose (Experimental): Participants received adavosertib 325 mg, orally, on Day 1.
  Interventions: Drug: adavosertib
- adavosertib 650 mg Single Dose (Experimental): Participants received adavosertib 650 mg, orally, on Day 1.
  Interventions: Drug: adavosertib
- adavosertib 1300 mg Single Dose (Experimental): Participants received adavosertib 1300 mg, orally, on Day 1.
  Interventions: Drug: adavosertib
- adavosertib 100 mg Single Dose + Gemcitabine 1000 mg/m^2 (Experimental): Participants received gemcitabine 1000 mg/m^2 as an intravenous (IV) infusion on Days 1, 8, and 15 in each 4-week cycle plus adavosertib 100 mg single dose, orally, on Day 2 of each cycle.
  Interventions: Drug: adavosertib; Drug: gemcitabine
- adavosertib 200 mg Single Dose + Gemcitabine 1000 mg/m^2 (Experimental): Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 in each 4-week cycle plus adavosertib 200 mg single dose, orally, on Day 2 of each cycle.
  Interventions: Drug: adavosertib; Drug: gemcitabine
- adavosertib 100 mg Single Dose + Cisplatin 75 mg/ m^2 (Experimental): Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 100 mg single dose orally, on Day 2 of each cycle.
  Interventions: Drug: adavosertib; Drug: cisplatin
- adavosertib 200 mg Single Dose + Cisplatin 75 mg/ m^2 (Experimental): Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 200 mg single dose orally, on Day 2 of each cycle.
  Interventions: Drug: adavosertib; Drug: cisplatin
- adavosertib 100 mg Single Dose + Carboplatin AUC 5 (Experimental): Participants received carboplatin at an area under the time curve concentration of 5 mg/min/ml (AUC5) as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 100 mg single dose orally, on Day 2 of each cycle.
  Interventions: Drug: adavosertib; Drug: carboplatin
- adavosertib 200 mg Single Dose + Carboplatin AUC 5 (Experimental): Participants received carboplatin AUC5 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 200 mg single dose orally, on Day 2 of each cycle.
  Interventions: Drug: adavosertib; Drug: carboplatin
- adavosertib 325 mg Single Dose + Carboplatin AUC 5 (Experimental): Participants received carboplatin AUC5 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 325 mg single dose orally, on Day 2 of each cycle.
  Interventions: Drug: adavosertib; Drug: carboplatin
- adavosertib 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2 (Experimental): Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4-week cycle plus adavosertib 25 mg orally twice daily (BID) for 2.5 days, starting concomitantly with the IV infusion of gemcitabine on Day 1 and followed by 4 additional doses of adavosertib 25 mg at approximately 12 hour intervals on Days 1-3, 8-9, and 15-17 of each cycle.
  Interventions: Drug: adavosertib; Drug: gemcitabine
- adavosertib 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 (Experimental): Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus adavosertib 50 mg orally BID for 2.5 days, starting concomitantly with the IV infusion of gemcitabine on Day 1 and followed by 4 doses of adavosertib 25 mg at approximately 12 hour intervals on Days 1-3, 8-9, and 15-17 of each 4 week cycle.
  Interventions: Drug: adavosertib; Drug: gemcitabine
- adavosertib 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 (Experimental): Participants received gemcitabine 1000 mg/m^2 as an IV infusion given once weekly for 3 consecutive weeks of a 4 week cycle plus adavosertib 50 mg orally BID for 2.5 days, starting concomitantly with the IV infusion of gemcitabine on Day 1 and followed by 4 additional doses of adavosertib 50 mg at approximately 12 hour intervals on Days 1-3, 8-9, and 15-17 of each 4 week cycle.
  Interventions: Drug: adavosertib; Drug: gemcitabine
- adavosertib 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 (Experimental): Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus adavosertib 100 mg orally once daily (QD) on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
  Interventions: Drug: adavosertib; Drug: gemcitabine
- adavosertib 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 (Experimental): Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus adavosertib 125 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
  Interventions: Drug: adavosertib; Drug: gemcitabine
- adavosertib 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 (Experimental): Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus adavosertib 150 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
  Interventions: Drug: adavosertib; Drug: gemcitabine
- adavosertib 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 (Experimental): Participants received gemcitabine 1000 mg/m^2 as an IV infusion given on Days 1, 8, and 15 of each 4 week cycle plus adavosertib 175 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
  Interventions: Drug: adavosertib; Drug: gemcitabine
- adavosertib 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 (Experimental): Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus adavosertib 200 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
  Interventions: Drug: adavosertib; Drug: gemcitabine
- adavosertib 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 (Experimental): Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 50 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
  Interventions: Drug: adavosertib; Drug: cisplatin
- adavosertib 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 (Experimental): Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 100 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
  Interventions: Drug: adavosertib; Drug: cisplatin
- adavosertib 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 (Experimental): Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 125 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
  Interventions: Drug: adavosertib; Drug: cisplatin
- adavosertib 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 (Experimental): Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 150 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
  Interventions: Drug: adavosertib; Drug: cisplatin
- adavosertib 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 (Experimental): Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 200 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
  Interventions: Drug: adavosertib; Drug: cisplatin
- adavosertib 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 (Experimental): Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 250 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
  Interventions: Drug: adavosertib; Drug: cisplatin
- adavosertib 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 (Experimental): Participants received carboplatin AUC 5 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 75 mg orally BID for 2.5 days, starting concomitantly with the administration of carboplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
  Interventions: Drug: adavosertib; Drug: carboplatin
- adavosertib 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5 (Experimental): Participants received carboplatin AUC 5 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 150 mg orally BID for 2.5 days, starting concomitantly with the administration of carboplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
  Interventions: Drug: adavosertib; Drug: carboplatin
- adavosertib 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 (Experimental): Participants received carboplatin AUC 5 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 225 mg orally BID for 2.5 days, starting concomitantly with the administration of carboplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
  Interventions: Drug: adavosertib; Drug: carboplatin
- adavosertib 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5 (Experimental): Participants received carboplatin AUC 5 as an IV infusion on Day 1 of each 3 week cycle plus adavosertib 325 mg orally BID for 2.5 days, starting concomitantly with the administration of carboplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
  Interventions: Drug: adavosertib; Drug: carboplatin

INTERVENTIONS:
Drug: adavosertib — adavosertib administered as an oral formulation as either monotherapy or in combination with either gemcitabine, cisplatin, or carboplatin.
  Other Names: MK-1775
Drug: gemcitabine — Gemcitabine administered at 1000 mg/m^2 by IV infusion in a 28-day cycle.
  Arms: adavosertib 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2; adavosertib 100 mg Single Dose + Gemcitabine 1000 mg/m^2; adavosertib 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2; adavosertib 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2; adavosertib 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2; adavosertib 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2; adavosertib 200 mg Single Dose + Gemcitabine 1000 mg/m^2; adavosertib 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2; adavosertib 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2; adavosertib 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2
Drug: cisplatin — Cisplatin administered at 75 mg/m^2 by IV infusion in a 21-day cycle.
  Arms: adavosertib 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2; adavosertib 100 mg Single Dose + Cisplatin 75 mg/ m^2; adavosertib 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2; adavosertib 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2; adavosertib 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2; adavosertib 200 mg Single Dose + Cisplatin 75 mg/ m^2; adavosertib 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2; adavosertib 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2
Drug: carboplatin — Carboplatin administered at AUC/time curve of 5 mg/min/mL (AUC5) by IV infusion in a 21-day cycle.
  Arms: adavosertib 100 mg Single Dose + Carboplatin AUC 5; adavosertib 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5; adavosertib 200 mg Single Dose + Carboplatin AUC 5; adavosertib 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5; adavosertib 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5; adavosertib 325 mg Single Dose + Carboplatin AUC 5; adavosertib 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5

SUMMARY:
This study will investigate the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) activity of adavosertib, both as monotherapy and in combination with gemcitabine, cisplatin, or carboplatin in participants with advanced solid tumors. Dose limiting toxicities (DLT) of adavosertib in combination with gemcitabine, cisplatin, or carboplatin will also be assessed. The primary hypotheses of the study are as follows: 1) Oral administration of adavosertib both as monotherapy and in combination with either gemcitabine, cisplatin, or carboplatin in patients with advanced solid tumors will be safe and tolerable, 2) The side effects observed in participants with advanced solid tumors after administration of adavosertib combined with each of the chemotherapies (gemcitabine, cisplatin and carboplatin) will allow for the definition of a single dose combination Maximum Administered Dose (MAD)/Maximum Tolerated Dose (MTD) and a multiple dose combination Biologically Effective Dose (BED)/MTD for each of the 3 combinations, 3) At a tolerated dose, adavosertib plasma exposure will exceed target thresholds established in preclinical models, and 4) At a tolerated dose, PD markers of adavosertib activity in combination with either gemcitabine, cisplatin, or carboplatin (in surrogate tissue and/or tumor) will meet or exceed the target threshold established in preclinical models.

DETAILED DESCRIPTION:
Part 1 consists of single dose adavosertib monotherapy. If well tolerated, participants in Part 1 will continue on to one of three treatment arms in Part 2-A which consists of a single lower dose of adavosertib in combination with standard chemotherapy: 1) Adavosertib +Gemcitabine (1000 mg/m^2), 2) Adavosertib + Cisplatin (75 mg/m^2) or 3) Adavosertib +Carboplatin at an area under the time curve concentration of 5 mg/min/ml (AUC5). Following completion of Part 2-A, adavosertib will be administered twice daily (BID) for 2.5 days (multi-dose) starting concomitantly with each administration of chemotherapy in Part 2-B. After a preliminary combination MTD of adavosertib and chemotherapy has been established in Part 2B, the MTD confirmation expansion will occur in Part 3.

ELIGIBILITY:
Inclusion Criteria:

* Must have a histologically confirmed metastatic or locally advanced solid tumor, progressed despite standard therapy, or for which standard therapy does not exist
* Must have performance status of <=1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Female participants must not be pregnant

Exclusion Criteria:

* Has had chemotherapy, radiotherapy, or biological therapy within 4 weeks prior to entering the study or who has not recovered from adverse events due to agents given more than 4 weeks earlier
* Is participating or has participated in a study with an investigational compound or device within 30 days
* Has active central nervous system (CNS) metastases and/or carcinomatous meningitis. However, participants with CNS metastases who have completed a course of therapy would be eligible for the study provided they are clinically stable for 1 month prior to entry
* Has a primary central nervous system tumor
* Is allergic to any of the components of the combination study therapy or its analogs
* Participant has had prescription or non-prescription drugs or other products known to be metabolized by Cytochrome P450 3A4 (CYP3A4) that cannot be discontinued prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study medication. Medications of particular concern are inhibitors of CYP3A4 (azole antifungals [ketoconazole, itraconazole], macrolide antibiotics [erythromycin, clarithromycin], cimetidine, aprepitant, Human Immunodeficiency Virus (HIV) protease inhibitors, nefrazodone, and the following inducers of CYP3A4: phenytoin, barbiturates and rifampicin, and substrates of CYP3A4 including statins (lovastatin, simvastatin), midazolam, terfenadine, astemizole, and cisapride
* Is a regular user (including "recreational use") of any illicit drugs or had a recent history (within the last year) of drug or alcohol abuse
* Pregnant or breastfeeding, or expecting to get pregnant during the time the study will be ongoing
* HIV-positive
* History of Hepatitis B or C
* Has symptomatic ascites or pleural effusion. A participant who is clinically stable following treatment for these conditions is eligible
* Participant must not have prior radiation therapy to more than 30% of the bone marrow and must have recovered for at least 3 weeks from the hematologic toxicity of prior radiotherapy
* Has had a prior stem cell or bone marrow transplant
* Has received more than 4 prior cytotoxic chemotherapy regimens
* Has a history suggestive of Li-Fraumeni Syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2008-02-25 (Actual); Primary Completion 2014-01-06 (Actual); Study Completion 2014-01-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Leijen S, van Geel RM, Pavlick AC, Tibes R, Rosen L, Razak AR, Lam R, Demuth T, Rose S, Lee MA, Freshwater T, Shumway S, Liang LW, Oza AM, Schellens JH, Shapiro GI. Phase I Study Evaluating WEE1 Inhibitor AZD1775 As Monotherapy and in Combination With Gemcitabine, Cisplatin, or Carboplatin in Patients With Advanced Solid Tumors. J Clin Oncol. 2016 Dec 20;34(36):4371-4380. doi: 10.1200/JCO.2016.67.5991. Epub 2016 Oct 31. PMID 27601554
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 206 participants were allocated to one of 28 treatment arms (3 Part 1 arms and 25 Part 2 arms). 8 participants from the Part 1 MK-1775 monotherapy arms continued into Part 2 of the study and received single dose (SD) combination treatment. For disposition purposes these participants are counted under Part 1 only.
Groups:
- MK-1775 325 mg Single Dose: Participants received MK-1775 325 mg, orally, on Day 1.
- MK-1775 650 mg Single Dose: Participants received MK-1775 650 mg, orally, on Day 1.
- MK-1775 1300 mg Single Dose: Participants received MK-1775 1300 mg, orally, on Day 1.
- MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m^2: Participants received gemcitabine 1000 mg/m^2 as an intravenous (IV) infusion on Days 1, 8, and 15 in each 4-week cycle plus MK-1775 100 mg single dose, orally, on Day 2 of each cycle.
- MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m^2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 in each 4-week cycle plus MK-1775 200 mg single dose, orally, on Day 2 of each cycle.
- MK-1775 100 mg Single Dose + Cisplatin 75 mg/ m^2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 100 mg single dose orally, on Day 2 of each cycle.
- MK-1775 200 mg Single Dose + Cisplatin 75 mg/ m^2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 200 mg single dose orally, on Day 2 of each cycle.
- MK-1775 100 mg Single Dose + Carboplatin AUC 5: Participants received carboplatin at an area under the time curve concentration of 5 mg/min/ml (AUC5) as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 100 mg single dose orally, on Day 2 of each cycle.
- MK-1775 200 mg Single Dose + Carboplatin AUC 5: Participants received carboplatin AUC5 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 200 mg single dose orally, on Day 2 of each cycle.
- MK-1775 325 mg Single Dose + Carboplatin AUC 5: Participants received carboplatin AUC5 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 325 mg single dose orally, on Day 2 of each cycle.
- MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4-week cycle plus MK-1775 25 mg orally twice daily (BID) for 2.5 days, starting concomitantly with the IV infusion of gemcitabine on Day 1 and followed by 4 additional doses of MK-1775 25 mg at approximately 12 hour intervals on Days 1-3, 8-9, and 15-17 of each cycle.
- MK-1775 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 50 mg orally BID for 2.5 days, starting concomitantly with the IV infusion of gemcitabine on Day 1 and followed by 4 doses of MK-1775 25 mg at approximately 12 hour intervals on Days 1-3, 8-9, and 15-17 of each 4 week cycle.
- MK-1775 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion given once weekly for 3 consecutive weeks of a 4 week cycle plus MK-1775 50 mg orally BID for 2.5 days, starting concomitantly with the IV infusion of gemcitabine on Day 1 and followed by 4 additional doses of MK-1775 50 mg at approximately 12 hour intervals on Days 1-3, 8-9, and 15-17 of each 4 week cycle.
- MK-1775 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 100 mg orally once daily (QD) on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
- MK-1775 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 125 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
- MK-1775 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 150 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
- MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion given on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 175 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
- MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 200 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
- MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 50 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 100 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 125 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 150 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 200 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 250 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5: Participants received carboplatin AUC 5 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 75 mg orally BID for 2.5 days, starting concomitantly with the administration of carboplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5: Participants received carboplatin AUC 5 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 150 mg orally BID for 2.5 days, starting concomitantly with the administration of carboplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5: Participants received carboplatin AUC 5 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 225 mg orally BID for 2.5 days, starting concomitantly with the administration of carboplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5: Participants received carboplatin AUC 5 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 325 mg orally BID for 2.5 days, starting concomitantly with the administration of carboplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
Period: Overall Study
Arm/Group | MK-1775 325 mg Single Dose | MK-1775 650 mg Single Dose | MK-1775 1300 mg Single Dose | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 100 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg Single Dose + Carboplatin AUC 5 | MK-1775 200 mg Single Dose + Carboplatin AUC 5 | MK-1775 325 mg Single Dose + Carboplatin AUC 5 | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5
Started (Started = Randomized) | 3 | 3 | 3 | 4 (Does not include two Part 1 participants who were randomized to this arm.) | 9 | 1 (Does not include two Part 1 participants who were randomized to this arm.) | 10 (Does not include one Part 1 participant who was randomized to this arm.) | 1 (Does not include two Part 1 participants who were randomized to this arm.) | 3 (Does not include one Part 1 participant who was randomized to this arm.) | 10 | 6 | 13 | 6 | 5 | 4 | 11 | 16 | 6 | 5 | 7 | 6 | 10 | 14 | 4 | 4 | 4 | 26 | 12
Treated | 3 | 3 | 3 | 4 (Does not include two Part 1 participants who were treated in this arm.) | 8 | 1 (Does not include two Part 1 participants who were treated in this arm.) | 9 (Does not include one treated participant who was excluded from analysis.) | 1 (Does not include two Part 1 participants who were treated in this arm.) | 3 (Does not include one Part 1 participant who was treated in this arm.) | 9 (Does not include one treated participant who was excluded from analysis.) | 6 | 13 | 6 | 5 | 4 | 11 | 16 | 6 | 4 | 7 | 6 | 10 | 14 | 4 | 4 | 4 | 26 | 12
Completed | 3 | 3 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 4 | 9 | 1 | 10 | 1 | 3 | 10 | 6 | 13 | 6 | 5 | 4 | 11 | 14 | 6 | 5 | 7 | 6 | 10 | 14 | 4 | 4 | 4 | 26 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-1775 325 mg Single Dose | MK-1775 650 mg Single Dose | MK-1775 1300 mg Single Dose | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 100 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg Single Dose + Carboplatin AUC 5 | MK-1775 200 mg Single Dose + Carboplatin AUC 5 | MK-1775 325 mg Single Dose + Carboplatin AUC 5 | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | Total
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 9 | 1 | 10 | 1 | 3 | 10 | 6 | 13 | 6 | 5 | 4 | 11 | 16 | 6 | 5 | 7 | 6 | 10 | 14 | 4 | 4 | 4 | 26 | 12 | 206
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.0 (13.7) | 44.0 (8.5) | 67.7 (19.5) | 47.0 (19.6) | 60.6 (12.6) | 58.0 (0) | 61.5 (10.2) | 75.0 (0) | 64.7 (4.0) | 55.6 (13.0) | 56.2 (6.8) | 55.1 (12.5) | 64.5 (10.7) | 49.8 (18.4) | 60.5 (8.3) | 64.7 (9.1) | 64.8 (8.9) | 57.8 (8.8) | 55.2 (7.5) | 56.1 (14.6) | 48.8 (12.4) | 51.5 (8.8) | 52.6 (9.4) | 62.3 (3.3) | 61.0 (9.6) | 65.8 (8.8) | 56.2 (12.8) | 58.5 (12.6) | 57.9 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8 | 0 | 4 | 0 | 0 | 5 | 3 | 10 | 3 | 3 | 1 | 5 | 11 | 3 | 3 | 2 | 3 | 5 | 10 | 4 | 2 | 2 | 14 | 7 | 116
  Male | 1 | 1 | 1 | 2 | 1 | 1 | 6 | 1 | 3 | 5 | 3 | 3 | 3 | 2 | 3 | 6 | 5 | 3 | 2 | 5 | 3 | 5 | 4 | 0 | 2 | 2 | 12 | 5 | 90

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Experiencing Dose-Limiting Toxicities (DLTs)
Description: DLTs were adverse events (AEs) considered at least possibly related to study drug that prevented escalation of the drug dose. Hematologic DLTs were any grade (Gr) 4-5 toxicity EXCEPT: Gr 4 anemia and Gr 4 leukopenia, Gr 4 neutropenia lasting for <7 days, Gr 4 thrombocytopenia lasting for <4 days except if a platelet transfusion is required, and Gr 3/Gr 4 neutropenia with fever >38.5°C and/or infection requiring antibiotic or anti-fungal treatment. Non-hematologic DLT was defined as any Gr 3, 4, or 5 non-hematologic toxicity EXCEPT: nausea, vomiting, diarrhea, or dehydration (all Gr 3) occurring in a setting of inadequate compliance with supportive care measures and lasting for <48 hours, alopecia of any grade, inadequately treated hypersensitivity reactions, and clinically non-significant, treatable or reversible lab abnormalities including liver function tests, uric acid, etc.
Time Frame: Part 1: Up to 14 days, Part 2: Up to 28 days
Population: All participants who received at least one dose of study treatment and were evaluable for DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1775 325 mg Single Dose | MK-1775 650 mg Single Dose | MK-1775 1300 mg Single Dose | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 100 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg Single Dose + Carboplatin AUC 5 | MK-1775 200 mg Single Dose + Carboplatin AUC 5 | MK-1775 325 mg Single Dose + Carboplatin AUC 5 | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 8 | 3 | 10 | 3 | 4 | 9 | 6 | 13 | 6 | 5 | 4 | 11 | 16 | 6 | 4 | 7 | 6 | 10 | 14 | 4 | 4 | 4 | 26 | 12
Participants | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 0 | 0 | 0 | 1 | 2 | 5 | 0 | 0 | 2 | 1 | 3 | 0 | 1 | 0 | 0 | 4 | 3 | 0 | 0 | 7 | 6

2. Primary Outcome: Percentage of Total Cyclin-dependent Kinase (CDC2)-Positive Cells That Were Phosphorylated (pCDC2) in Skin Cells at Baseline and 8 Hours After MK-1775 Dosing
Description: The pCDC2 level in skin cells was used as a marker to evaluate MK-1775 activity. Analysis was done by immunohistochemistry and the percentage of total CDC2-positive cells that were pCDC2 positive (% pCDC2-positive cells) at baseline and 8 hours after MK-1775 dosing were reported for participants in Part 1, 2-A, and 2-B/3 treatment groups with available data per protocol.
Time Frame: Baseline, 8 hours after first MK-1775 dose
Population: Participants in Parts 1, 2-A, and 2-B/3 with ≥1 dose treatment and evaluable CDC2 data at 8 hours post dosing. Per protocol the MK-1775 QD x2.5 Multi Dose + Gemcitabine groups, MK-1775 150, 200, and 250 mg BID x 2.5 Multi Dose + cisplatin 75 mg/m^2 groups, and MK-1775 325 mg BID x 2.5 Multi Dose + carboplatin AUC 5 group did not have data reported
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: percentage of cells
Arm/Group | MK-1775 325 mg Single Dose | MK-1775 650 mg Single Dose | MK-1775 1300 mg Single Dose | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 100 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg Single Dose + Carboplatin AUC 5 | MK-1775 200 mg Single Dose + Carboplatin AUC 5 | MK-1775 325 mg Single Dose + Carboplatin AUC 5 | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5
Number analyzed (Participants) | 3 | 3 | 3 | 4 | 7 | 1 | 9 | 1 | 3 | 8 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 1 | 0 | 0 | 0 | 4 | 4 | 8 | 0
percentage of cells
  Baseline percentage: number analyzed (Participants) | 3 | 3 | 3 | 4 | 7 | 1 | 9 | 1 | 3 | 7 | 6 | 6 | 6 | 0 | 0 | 0 | 0 | 0 | 3 | 7 | 1 | 0 | 0 | 0 | 4 | 4 | 8 | 0
  Baseline percentage | 40.8 [26.6 to 62.7] | 35.1 [22.8 to 54] | 36.2 [23.6 to 55.7] | 53.2 [36.7 to 77.2] | 40.7 [30.7 to 53.9] | 16.1 [7.6 to 33.8] | 28.6 [22.3 to 36.7] | 34.4 [16.3 to 72.4] | 17.6 [11.4 to 27] | 22.4 [17 to 29.6] | 28.1 [20.7 to 38.1] | 18.3 [13.5 to 24.8] | 30.8 [22.7 to 41.7] |  |  |  |  |  | 16.4 [10.7 to 25.2] | 24.1 [18.2 to 31.9] | 21.4 [10.2 to 45.1] |  |  |  | 15.7 [10.9 to 22.8] | 27 [18.6 to 39.2] | 21 [15.9 to 27.8] |
  Percentage after dosing | 18 [9.3 to 34.7] | 13.4 [6.9 to 25.8] | 20.6 [10.7 to 39.9] | 28.9 [16.3 to 51.2] | 35.7 [23.2 to 55] | 14.8 [4.7 to 46.4] | 22.1 [15.1 to 32.4] | 41.9 [13.4 to 131.3] | 20.9 [10.8 to 40.3] | 17.1 [11.4 to 25.6] | 20.1 [12.6 to 32] | 13.7 [8.6 to 21.8] | 16.6 [10.4 to 26.4] |  |  |  |  |  | 17.8 [9.2 to 34.4] | 14.4 [9.3 to 22.1] | 19.9 [6.3 to 62.2] |  |  |  | 12.1 [6.9 to 21.5] | 16.8 [9.5 to 29.6] | 11.5 [7.7 to 17.2] |

3. Primary Outcome: Percentage of Total pCDC2 in Skin Cells at Baseline and 24 Hours After MK-1775 Dosing
Description: The pCDC2 level in skin cells was used as a marker to evaluate MK-1775 activity. Analysis was done by immunohistochemistry and the percentage of total pCDC2 at baseline and 24 hours after MK-1775 dosing were reported for participants in the Part 2-B/3 MK-1775 QD x2 Multi Dose plus Gemcitabine treatment groups with available data per protocol.
Time Frame: Baseline, 24 hours after first MK-1775 dose
Population: All participants in the Part 2-B/3 MK-1775 QD x2 Multi Dose plus Gemcitabine treatment groups who received at least one dose of study treatment and had evaluable CDC2 data at 24 hours post dosing. Per protocol, the Part 1, Part 2-A, and Part 2-B/3 MK-1775 BID treatment groups did not have data reported for this time point.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: percentage of cells
Arm/Group | MK-1775 325 mg Single Dose | MK-1775 650 mg Single Dose | MK-1775 1300 mg Single Dose | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 100 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg Single Dose + Carboplatin AUC 5 | MK-1775 200 mg Single Dose + Carboplatin AUC 5 | MK-1775 325 mg Single Dose + Carboplatin AUC 5 | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 4 | 11 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
percentage of cells
  Baseline percentage |  |  |  |  |  |  |  |  |  |  |  |  |  | 47.5 [32.6 to 69.2] | 27.9 [19.1 to 40.7] | 18.7 [14.9 to 23.5] |  | 11.6 [7.9 to 16.9] |  |  |  |  |  |  |  |  |  |
  Percentage after dosing |  |  |  |  |  |  |  |  |  |  |  |  |  | 29.9 [17.3 to 51.9] | 17.7 [10.2 to 30.7] | 12.7 [9.1 to 17.7] |  | 6.3 [3.6 to 11] |  |  |  |  |  |  |  |  |  |

4. Primary Outcome: Percentage of Total pCDC2 in Skin Cells at Baseline and 48 Hours After MK-1775 Dosing
Description: The pCDC2 level in skin cells was used as a marker to evaluate MK-1775 activity. Analysis was done by immunohistochemistry and the percentage of total pCDC2 at baseline and at 48 hours after MK-1775 dosing were reported for participants in the Part 2-B/3 MK-1775 (150 mg, 200 mg, 250) BID x 2.5 Multi Dose plus cisplatin 75 mg/m^2 groups and the 325 mg BID x2.5 Multi Dose + Carboplatin group with available data per protocol.
Time Frame: Baseline, 48 hours after first MK-1775 dose
Population: All participants in Part 2-B/3 MK-1775 (150 mg, 200 mg, 250) BID x 2.5 Multi Dose plus cisplatin 75 mg/m^2 groups and 325 mg BID x2.5 Multi Dose + carboplatin group who received ≥1 dose of study treatment and had evaluable CDC2 data at 48 hours post dose. Per protocol, Part 1, Part 2-A, and remaining Part 2-B/3 groups did not have data reported.
Measure: Geometric Least Squares Mean (90% Confidence Interval); unit: percentage of cells
Arm/Group | MK-1775 325 mg Single Dose | MK-1775 650 mg Single Dose | MK-1775 1300 mg Single Dose | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 100 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg Single Dose + Carboplatin AUC 5 | MK-1775 200 mg Single Dose + Carboplatin AUC 5 | MK-1775 325 mg Single Dose + Carboplatin AUC 5 | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 8 | 9 | 4 | 0 | 0 | 0 | 9
percentage of cells
  Baseline percentage |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 28.6 [23.6 to 34.6] | 31.5 [26.3 to 37.8] | 31.5 [24 to 41.3] |  |  |  | 33.5 [28 to 40.2]
  Percentage after dosing |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  | 15.7 [10 to 24.8] | 7.4 [4.8 to 11.4] | 11.1 [5.9 to 21.1] |  |  |  | 15.1 [9.8 to 23.1]

5. Primary Outcome: Plasma Concentration of MK-1775 at 8 Hours After Administration (C8hr) of Single or Multiple Oral Doses
Description: MK-1775 was measured in the plasma at 8 hours after dosing (Day 1 for single dose of monotherapy, Day 2 of single-dose combination therapy and QD x 2 Combination dosing, and Day 3 dose for BID X 2.5 combination dosing) for participants with available data.
Time Frame: 8 hours after MK-1775 dose
Population: All treated participants with available C8hr data.
Measure: Mean (Standard Deviation); unit: nM
Arm/Group | MK-1775 325 mg Single Dose | MK-1775 650 mg Single Dose | MK-1775 1300 mg Single Dose | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 100 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg Single Dose + Carboplatin AUC 5 | MK-1775 200 mg Single Dose + Carboplatin AUC 5 | MK-1775 325 mg Single Dose + Carboplatin AUC 5 | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5
Number analyzed (Participants) | 3 | 3 | 3 | 6 | 7 | 3 | 8 | 2 | 4 | 8 | 6 | 13 | 5 | 4 | 3 | 11 | 11 | 6 | 4 | 7 | 5 | 7 | 10 | 3 | 4 | 4 | 13 | 11
nM | 585 (262) | 1130 (73.2) | 2190 (791) | 129 (46.5) | 235 (136) | 108 (62.7) | 310 (168) | 119 (0.706) | 262 (52.1) | 425 (190) | 41.7 (16.3) | 65.4 (26.1) | 138 (38.8) | 188 (47.6) | 241 (92.3) | 355 (230) | 346 (144) | 407 (183) | 113 (97.7) | 388 (149) | 748 (234) | 920 (439) | 1070 (528) | 2010 (581) | 184 (101) | 295 (161) | 985 (301) | 1960 (651)

6. Primary Outcome: Mean Urine Excretion of MK-1775 24 Hours After the Day 1 Monotherapy Dose
Description: The mean cumulative amount of MK-1775 excreted unchanged in urine after a single oral dose was measured during the initial monotherapy cycle of the study. For this outcome measure, samples were collected and analyzed only for the MK-1775 monotherapy arms of the study at defined intervals after the Day 1 dose of monotherapy. Part 2 MK-1775 combination arms were not sampled per protocol.
Time Frame: At 0-4 hours, 4-8 hours, and 12-24 hours post Day 1 dose of monotherapy
Population: All treated Part 1 participants with available urine sample data.
Measure: Mean (Standard Deviation); unit: mg
Arm/Group | MK-1775 325 mg Single Dose | MK-1775 650 mg Single Dose | MK-1775 1300 mg Single Dose | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 100 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg Single Dose + Carboplatin AUC 5 | MK-1775 200 mg Single Dose + Carboplatin AUC 5 | MK-1775 325 mg Single Dose + Carboplatin AUC 5 | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5
Number analyzed (Participants) | 1 | 3 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
mg | 16.7 (NA) — Standard Deviation not calculated since n=1 | 35.4 (9.86) | 154 (NA) — Standard Deviation not calculated since n=1 |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |  |

7. Secondary Outcome: Best Overall Response as Per Response Evaluation Criteria in Solid Tumors (RECIST) Criteria
Description: Best overall response achieved by a participant. Starting at Day 1, participants in Part 2 were evaluated for tumor response every 6-8 weeks until discontinuation from study treatment according to RECIST criteria; which are based on radiographic imaging. Recorded responses were either confirmed by Central Review or unconfirmed (Investigator assessment only), and included complete response (CR; defined as disappearance of all target lesions), partial response (PR; at least a 30% decrease in the sum of the longest diameter [LD] of target lesions, taking as reference the baseline sum LD), stable disease (SD; neither sufficient shrinkage to qualify for PR nor sufficient growth to qualify for PD, taking as reference the smallest sum LD since the treatment started), or progressive disease (PD; ≥20% increase in sum of the LD of target lesions, taking as reference the smallest sum LD recorded since the treatment started, or the appearance of one or more new lesions).
Time Frame: From Day 1 up through discontinuation of study treatment (up to ~11.2 months)
Population: All treated participants in Part 2 with measurable disease at baseline per RECIST criteria. Participants who were originally treated in Part 1 and continued in Part 2 were included in their respective Part 2 arms. Participants who could not be evaluated after treatment are categorized as "not evaluable (NE).
Measure: Count of Participants; unit: Participants
Arm/Group | MK-1775 325 mg Single Dose | MK-1775 650 mg Single Dose | MK-1775 1300 mg Single Dose | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m^2 | MK-1775 100 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg Single Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg Single Dose + Carboplatin AUC 5 | MK-1775 200 mg Single Dose + Carboplatin AUC 5 | MK-1775 325 mg Single Dose + Carboplatin AUC 5 | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50/25 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 100 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 125 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 150 mg QD x2 Multi + Gemcitabine 1000 mg/ m^2 | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/ m^2 | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/ m^2 | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 150 mg BID x 2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5
Number analyzed (Participants) | 0 | 0 | 0 | 6 | 6 | 3 | 9 | 3 | 3 | 9 | 5 | 9 | 5 | 4 | 4 | 10 | 13 | 5 | 3 | 5 | 5 | 10 | 11 | 4 | 4 | 4 | 24 | 12
Participants
  CR | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Confirmed PR | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  Unconfirmed PR | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 2 | 0
  SD | 0 | 0 | 0 | 3 | 5 | 0 | 7 | 0 | 0 | 3 | 4 | 4 | 4 | 2 | 2 | 8 | 8 | 3 | 2 | 1 | 1 | 4 | 6 | 2 | 2 | 3 | 14 | 6
  PD | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 3 | 3 | 3 | 1 | 5 | 1 | 2 | 2 | 2 | 3 | 1 | 1 | 2 | 4 | 4 | 3 | 1 | 2 | 1 | 8 | 6
  NE | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 30 days after the last dose of study drug (up to ~11.7 months)
Description: All participants receiving at least one dose of study medication.
Groups:
- MK-1775 650 mg Single Dose: Participants received MK-1775 650 mg, orally
- MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m2: Participants received gemcitabine 1000 mg/m^2 as an intravenous (IV) infusion on Days 1, 8, and 15 in each 4-week cycle plus MK-1775 100 mg single dose, orally, on Day 2 of each cycle.
- MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 in each 4-week cycle plus MK-1775 200 mg single dose, orally, on Day 2 of each cycle.
- MK-1775 100 mg Single Dose + Cisplatin 75 mg/m2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 100 mg single dose orally, on Day 2 of each cycle.
- MK-1775 200 mg Single Dose + Cisplatin 75 mg/m2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 200 mg single dose orally, on Day 2 of each cycle.
- MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4-week cycle plus MK-1775 25 mg orally twice daily (BID) for 2.5 days, starting concomitantly with the IV infusion of gemcitabine on Day 1 and followed by 4 additional doses of MK-1775 25 mg at approximately 12 hour intervals on Days 1-3, 8-9, and 15-17 of each cycle.
- MK-1775 50/25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 50 mg orally BID for 2.5 days, starting concomitantly with the IV infusion of gemcitabine on Day 1 and followed by 4 doses of MK-1775 25 mg at approximately 12 hour intervals on Days 1-3, 8-9, and 15-17 of each 4 week cycle.
- MK-1775 50 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion given once weekly for 3 consecutive weeks of a 4 week cycle plus MK-1775 50 mg orally BID for 2.5 days, starting concomitantly with the IV infusion of gemcitabine on Day 1 and followed by 4 additional doses of MK-1775 50 mg at approximately 12 hour intervals on Days 1-3, 8-9, and 15-17 of each 4 week cycle.
- MK-1775 100 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 100 mg orally once daily (QD) on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
- MK-1775 125 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 125 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
- MK-1775 150 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 150 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
- MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion given on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 175 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
- MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2: Participants received gemcitabine 1000 mg/m^2 as an IV infusion on Days 1, 8, and 15 of each 4 week cycle plus MK-1775 200 mg orally QD on Days 1, 2, 8, 9, 15, and 16 of each 4 week cycle.
- MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 50 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 100 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 125 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 150 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 200 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2: Participants received cisplatin 75 mg/ m^2 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 250 mg orally BID for 2.5 days, starting concomitantly with the administration of cisplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
- MK-1775 150 mg BID x2.5 Multi Dose + Carboplatin AUC 5: Participants received carboplatin AUC 5 as an IV infusion on Day 1 of each 3 week cycle plus MK-1775 150 mg orally BID for 2.5 days, starting concomitantly with the administration of carboplatin on Day 1 and then at 12 hour intervals on Days 1-3 of each 3 week cycle.
Arm/Group | MK-1775 325 mg Single Dose | MK-1775 650 mg Single Dose | MK-1775 1300 mg Single Dose | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m2 | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m2 | MK-1775 100 mg Single Dose + Cisplatin 75 mg/m2 | MK-1775 200 mg Single Dose + Cisplatin 75 mg/m2 | MK-1775 100 mg Single Dose + Carboplatin AUC 5 | MK-1775 200 mg Single Dose + Carboplatin AUC 5 | MK-1775 325 mg Single Dose + Carboplatin AUC 5 | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2 | MK-1775 50/25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2 | MK-1775 50 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2 | MK-1775 100 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 | MK-1775 125 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 | MK-1775 150 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 150 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 0/6 | 1/8 | 0/3 | 0/10 | 0/3 | 0/4 | 0/9 | 1/6 | 2/13 | 0/6 | 0/5 | 1/4 | 0/11 | 0/16 | 1/6 | 0/4 | 0/7 | 0/6 | 0/10 | 2/14 | 0/4 | 0/4 | 0/4 | 0/26 | 1/12
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3 | 0/3 | 1/6 | 3/8 | 1/3 | 3/10 | 1/3 | 1/4 | 1/9 | 3/6 | 6/13 | 0/6 | 2/5 | 3/4 | 4/11 | 4/16 | 5/6 | 1/4 | 0/7 | 3/6 | 5/10 | 6/14 | 2/4 | 1/4 | 0/4 | 13/26 | 7/12
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3 | 1/3 | 6/6 | 8/8 | 3/3 | 10/10 | 3/3 | 2/4 | 9/9 | 6/6 | 13/13 | 6/6 | 5/5 | 4/4 | 11/11 | 16/16 | 6/6 | 4/4 | 7/7 | 6/6 | 10/10 | 13/14 | 4/4 | 4/4 | 4/4 | 26/26 | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1775 325 mg Single Dose (N=3) | MK-1775 650 mg Single Dose (N=3) | MK-1775 1300 mg Single Dose (N=3) | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m2 (N=6) | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m2 (N=8) | MK-1775 100 mg Single Dose + Cisplatin 75 mg/m2 (N=3) | MK-1775 200 mg Single Dose + Cisplatin 75 mg/m2 (N=10) | MK-1775 100 mg Single Dose + Carboplatin AUC 5 (N=3) | MK-1775 200 mg Single Dose + Carboplatin AUC 5 (N=4) | MK-1775 325 mg Single Dose + Carboplatin AUC 5 (N=9) | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2 (N=6) | MK-1775 50/25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2 (N=13) | MK-1775 50 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2 (N=6) | MK-1775 100 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 (N=5) | MK-1775 125 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 (N=4) | MK-1775 150 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 (N=11) | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 (N=16) | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 (N=6) | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=4) | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=7) | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=6) | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=10) | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=14) | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=4) | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 (N=4) | MK-1775 150 mg BID x2.5 Multi Dose + Carboplatin AUC 5 (N=4) | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 (N=26) | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5 (N=12)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Faecaloma (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Asthenia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drug withdrawal syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Recall phenomenon (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Electrocardiogram ST-T segment elevation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal cord compression (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhage (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombophlebitis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-1775 325 mg Single Dose (N=3) | MK-1775 650 mg Single Dose (N=3) | MK-1775 1300 mg Single Dose (N=3) | MK-1775 100 mg Single Dose + Gemcitabine 1000 mg/m2 (N=6) | MK-1775 200 mg Single Dose + Gemcitabine 1000 mg/m2 (N=8) | MK-1775 100 mg Single Dose + Cisplatin 75 mg/m2 (N=3) | MK-1775 200 mg Single Dose + Cisplatin 75 mg/m2 (N=10) | MK-1775 100 mg Single Dose + Carboplatin AUC 5 (N=3) | MK-1775 200 mg Single Dose + Carboplatin AUC 5 (N=4) | MK-1775 325 mg Single Dose + Carboplatin AUC 5 (N=9) | MK-1775 25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2 (N=6) | MK-1775 50/25 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2 (N=13) | MK-1775 50 mg BID x2.5 Multi Dose + Gemcitabine 1000 mg/m2 (N=6) | MK-1775 100 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 (N=5) | MK-1775 125 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 (N=4) | MK-1775 150 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 (N=11) | MK-1775 175 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 (N=16) | MK-1775 200 mg QD x2 Multi Dose + Gemcitabine 1000 mg/m2 (N=6) | MK-1775 50 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=4) | MK-1775 100 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=7) | MK-1775 125 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=6) | MK-1775 150 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=10) | MK-1775 200 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=14) | MK-1775 250 mg BID x2.5 Multi Dose + Cisplatin 75 mg/m2 (N=4) | MK-1775 75 mg BID x2.5 Multi Dose + Carboplatin AUC 5 (N=4) | MK-1775 150 mg BID x2.5 Multi Dose + Carboplatin AUC 5 (N=4) | MK-1775 225 mg BID x2.5 Multi Dose + Carboplatin AUC 5 (N=26) | MK-1775 325 mg BID x2.5 Multi Dose + Carboplatin AUC 5 (N=12)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 2 (7) | 4 (4) | 0 (0) | 3 (5) | 1 (1) | 0 (0) | 4 (6) | 4 (11) | 9 (15) | 2 (4) | 1 (9) | 1 (1) | 8 (18) | 3 (4) | 2 (5) | 0 (0) | 0 (0) | 2 (3) | 4 (5) | 3 (4) | 2 (4) | 1 (1) | 0 (0) | 13 (25) | 5 (18)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 (0) | 4 (5) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (5) | 2 (4) | 3 (4) | 1 (3) | 1 (1) | 1 (1) | 3 (6) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 3 (9) | 3 (8)
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (3) | 3 (4) | 1 (1) | 3 (6) | 0 (0) | 0 (0) | 2 (7) | 2 (2) | 1 (1) | 4 (18) | 0 (0) | 1 (1) | 7 (21) | 10 (20) | 4 (6) | 0 (0) | 3 (4) | 0 (0) | 4 (4) | 4 (10) | 1 (1) | 1 (1) | 0 (0) | 10 (14) | 5 (14)
Pancytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 5 (12) | 3 (8) | 8 (16) | 4 (14) | 2 (7) | 3 (13) | 8 (34) | 9 (21) | 4 (7) | 0 (0) | 1 (1) | 2 (2) | 3 (3) | 5 (18) | 4 (12) | 1 (1) | 1 (2) | 19 (53) | 6 (25)
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Supraventricular extrasystoles (Cardiac disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cerumen impaction (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness bilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Ear congestion (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
External ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (5) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Deposit eye (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diplopia (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye discharge (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Eye swelling (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lacrimation increased (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ophthalmoplegia (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photophobia (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Photopsia (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vision blurred (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Visual impairment (Eye disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (5)
Abdominal hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 3 (4) | 1 (2) | 0 (0) | 2 (5) | 0 (0) | 5 (7) | 2 (5) | 2 (2) | 0 (0) | 1 (1) | 3 (3) | 3 (6) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (6)
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Anal fissure (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anorectal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chapped lips (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis ischaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 3 (3) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 3 (6) | 1 (1) | 6 (6) | 2 (3) | 2 (2) | 3 (3) | 2 (10) | 6 (10) | 3 (8) | 3 (6) | 3 (4) | 0 (0) | 8 (14) | 7 (10) | 1 (2) | 0 (0) | 1 (3) | 13 (24) | 3 (6)
Diarrhoea (Gastrointestinal disorders) | 0 | 2 (2) | 0 | 1 (1) | 2 (4) | 1 (1) | 5 (8) | 1 (1) | 1 (1) | 3 (4) | 2 (3) | 5 (6) | 5 (8) | 2 (3) | 1 (1) | 5 (7) | 5 (7) | 4 (8) | 1 (2) | 3 (13) | 2 (2) | 6 (12) | 6 (14) | 3 (3) | 2 (2) | 3 (4) | 18 (47) | 11 (20)
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Duodenitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 5 (10) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperchlorhydria (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melaena (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 | 0 | 4 (7) | 5 (13) | 1 (3) | 8 (14) | 1 (1) | 1 (1) | 5 (11) | 4 (14) | 7 (14) | 4 (5) | 4 (8) | 4 (6) | 9 (15) | 9 (15) | 4 (11) | 4 (9) | 6 (13) | 6 (10) | 10 (25) | 12 (46) | 4 (8) | 3 (4) | 3 (11) | 17 (38) | 8 (20)
Oesophageal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral pruritus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Retching (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 1 (1) | 3 (4) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 4 (6) | 3 (3)
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 (2) | 4 (10) | 1 (1) | 5 (9) | 0 (0) | 1 (1) | 2 (4) | 1 (10) | 3 (4) | 1 (1) | 2 (3) | 2 (3) | 3 (4) | 4 (4) | 4 (8) | 2 (2) | 5 (9) | 1 (1) | 6 (15) | 8 (13) | 3 (3) | 3 (3) | 3 (5) | 11 (15) | 7 (14)
Asthenia (General disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Axillary pain (General disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chest pain (General disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1)
Chills (General disorders) | 0 | 0 | 0 | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 1 (2) | 1 (3) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (3)
Face oedema (General disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 | 1 (1) | 1 (1) | 5 (12) | 5 (7) | 2 (2) | 6 (13) | 2 (2) | 1 (1) | 4 (7) | 6 (18) | 6 (10) | 4 (11) | 3 (4) | 3 (6) | 6 (20) | 10 (15) | 5 (14) | 3 (7) | 5 (9) | 3 (3) | 8 (11) | 8 (29) | 3 (5) | 2 (3) | 3 (6) | 18 (40) | 7 (15)
Feeling cold (General disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hernia pain (General disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 | 1 (1) | 0 | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (5) | 1 (1) | 3 (4) | 0 (0) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Local swelling (General disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised oedema (General disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 | 0 | 0 | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 4 (5) | 5 (6)
Mucosal inflammation (General disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 6 (6) | 3 (3) | 1 (1) | 1 (3) | 2 (2) | 2 (2) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (4) | 0 (0) | 0 (0) | 1 (3) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 | 1 (1) | 0 | 3 (7) | 3 (5) | 2 (2) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 2 (13) | 3 (10) | 5 (14) | 1 (2) | 3 (5) | 5 (9) | 4 (10) | 4 (9) | 1 (1) | 1 (1) | 4 (5) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 8 (11) | 2 (4)
Hepatic pain (Hepatobiliary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 | 0 | 0 | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 1 (1) | 3 (8) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Diverticulitis (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal infection (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes virus infection (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 | 1 (1) | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (2)
Oral candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Periodontitis (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Postoperative wound infection (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin infection (Infections and infestations) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection (Infections and infestations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Excoriation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Periorbital haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Postoperative wound complication (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase decreased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (10) | 1 (1) | 1 (6) | 3 (3) | 2 (2) | 1 (2) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (8) | 1 (6) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase decreased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 0 | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (7) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (3) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Blood bicarbonate decreased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood creatinine increased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (3) | 4 (12) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body temperature increased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphocyte count decreased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (7) | 0 (0) | 0 (0) | 1 (1) | 1 (4)
Platelet count decreased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Weight decreased (Investigations) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 4 (4) | 3 (4) | 1 (1) | 2 (2) | 3 (3) | 3 (3) | 3 (4) | 2 (2) | 3 (5) | 2 (2) | 2 (2) | 3 (5) | 1 (1) | 0 (0) | 1 (1) | 6 (7) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (3) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 1 (4) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 4 (5) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 4 (4) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 2 (2) | 2 (4)
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (3) | 2 (5) | 0 (0) | 0 (0) | 1 (7) | 2 (3)
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 1 (3)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 (1) | 0 | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 1 (4) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 3 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Finger deformity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Limb discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 1 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (7) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (6) | 3 (3) | 2 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amnesia (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Asterixis (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Burning sensation (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cognitive disorder (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 | 0 | 2 (2) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 2 (2) | 1 (2) | 1 (1) | 4 (6) | 4 (4)
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Head discomfort (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (6) | 2 (3) | 1 (2) | 1 (2) | 3 (15) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 2 (2) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 4 (4) | 2 (3)
Horner's syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 6 (7) | 4 (5)
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Delusion (Psychiatric disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephropathy (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurogenic bladder (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nocturia (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urinary hesitation (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal oedema (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scrotal swelling (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 2 (2) | 1 (2) | 1 (1) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 5 (6) | 4 (4)
Diaphragmalgia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 2 (2) | 4 (6) | 0 (0) | 1 (1) | 3 (3) | 2 (2) | 2 (2) | 1 (1) | 3 (3) | 2 (3) | 2 (2) | 1 (1) | 2 (2) | 3 (3) | 3 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 3 (4) | 6 (6) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Blister (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Plantar erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 3 (3) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 2 (2) | 3 (3) | 2 (7) | 1 (1) | 2 (2) | 3 (6) | 5 (6) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 3 (4) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (6) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin discolouration (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hot flush (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Intra-abdominal haematoma (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphoedema (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral vascular disorder (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Phlebitis (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The SPONSOR must have the opportunity to review all proposed abstracts, manuscripts, or presentations regarding this study 60 days prior to submission for publication/presentation. Any information identified by the SPONSOR as confidential must be deleted prior to submission. SPONSOR review can be expedited to meet publication timelines.